CLINICAL TRIAL: NCT01259765
Title: Safety and Tolerability of a Novel Llama-derived Anti-rotavirus VHH Fragment in Human Volunteers (Part-I), and Its Effect on Severity and Duration of Rotavirus Diarrhoea in Children (Part II). (This Registration Only Covers Part II)
Brief Title: Llama Antibody, Rotavirus Diarrhoea, Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Unilever Nederland Holdings (Unknown)
Responsible Party: Dr.Shafiqul Alam Sarker, International Centre for Diarrhoeal Disease Research, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004-009
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2006-02

CONDITIONS: Male Children; 6-24 Months Old With Rotaviral Diarrhoea; Non-cholera Patients
Keywords: llama antibody; rotavirus diarrhoea; children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VHH (Active Comparator): The active substance is "VHH batch 203027".
  Interventions: Drug: VHH batch 203027
- Placebo (Placebo Comparator): Placebo product
  Interventions: Drug: Placebo product

INTERVENTIONS:
Drug: VHH batch 203027 — The active product is 165 mg of VHH batch 203027 and 835 mg maltodextrin with 0.5% (w/w) caramel colour in 10 mL ORS. The osmolality (concentration of the osmotically active substances in the solution such as sugar molecules, salts etc. ) of this solution will be around 60 mOsmol/kg. The mixture of the 165 mg of VHH batch 203027 and 835 mg maltodextrin (0.5% (w/w) caramel colour will be provided per sachet.
  Arms: VHH
Drug: Placebo product — The Placebo treatment consisted of 1000 mg of maltodextrine with 5% (w/w) caramel colour in 10 mL ORS.
  Arms: Placebo

SUMMARY:
The investigators hypothesize that :

oral administration of VHH batch 203027 will be

* safe and tolerable for healthy Bangladeshi humans of all age groups (Part I)
* effective in reducing severity of diarrhoea in children with proven rotavirus infection (Part II). This entry only covers Part II.

DETAILED DESCRIPTION:
Brief Summary Study investigating the efficacy of oral administration of VHH antibody fragment derived from antibodies as found in milk of llamas and camels via a prototype food product in reducing the severity of rotavirus diarrhoea in children.

Detailed Description

Introduction Rotavirus is the leading viral enteropathogen, which is responsible for 11-71% of all diarrhoea episodes in infants and children worldwide. In developing countries, rotavirus is associated with more than 125 million episodes of diarrhoea each year (Cook et al. 1990), leading to an estimated 600,000 deaths. It is responsible for 60% of all diarrhoeal episodes, 20-60% of diarrhoeal hospitalizations, and 20% of diarrhoea-related deaths in children <5 years of age (Perez-Schael et al. 1997). In the United States of America alone, rotavirus is associated with 3% of all hospitalizations of children younger than 5 years with medical and indirect costs of over US$ 1 billion each year (Glass et al. 1991). In many localities deaths from rotavirus infections persist despite national programs to encourage the use of oral rehydration therapy.

Current management of rotavirus gastroenteritis Current management of rotavirus diarrhoea includes prevention of dehydration, or management of dehydration using oral or intravenous rehydration, as appropriate, and continued feeding. Early resumption of normal feeding is encouraged to enhance mucosal repair and to minimize nutritional consequences of infection. The children of developing countries might benefit from zinc supplementation, but its mode of delivery and cost effectiveness are yet to be decided in rotavirus diarrhoea. No specific treatment is currently available to reduce the duration or severity of this illness. Therefore, rotavirus-induced diarrhoea, which is considered to be a self-limited disease, is responsible for significant childhood deaths in the developing countries (Glass et al. 1996).

Active immunization against rotavirus infection The development, testing and eventual use of an effective, safe and inexpensive rotavirus vaccine would be the most efficient method for preventing severe disease and deaths in developing countries. Rapid progress has been made, and several candidate rotavirus vaccines have been developed and tested. Two rotavirus vaccines, Rotarix (GlaxoSmithKline Biologicals, Belgium) and RotaTeq (Merck & Co., USA) have recently entered the market in the developed world. Both vaccines appear to be safe with respect to intussusception, and are highly efficacious in preventing severe gastroenteritis due to rotavirus strains carrying predominantly serotype G1 (Cunliffe & Nakagomi 2005). Confirmation of the safety and efficacy of both vaccines in developing countries is still needed. Moreover, assessment of the ability of each vaccine to provide protection against increasingly diverse population of rotavirus strains will depend on continuous surveillance on the strain and development of newer vaccines as newer serotypes predominate in different geographical locations, which may not be easy for the developing countries. There thus is a clear need to define improved, cost effective interventions in the management of rotavirus diarrhoea until the time an effective, safe and inexpensive vaccine, affordable to the developing countries, is available.

Passive immunisation for rotavirus-induced diarrhoea; There are good reasons to hypothesize that passive immunisation could be useful in the management of human rotavirus diarrhoea. For example, oral administration of rotavirus-neutralizing antibodies has been found to modulate the rotavirus-induced diarrhoea in children. Beneficial prophylactic (Barnes et al. 1982) and therapeutic effects (Guarino et al. 1991), in terms of reduction of duration and severity of rotavirus diarrhoea, have also been observed in association with orally administered human IgG preparations. The use of human antibody preparation, however, is limited due to the risk of viral contamination and high production and supply chain costs of such product(s) and very low bio-availability.

An alternative source of antibodies, safe and easy to produce, was later developed in hyper immunized bovine colostrums by vaccinating pregnant cows against human strains of rotavirus. This approach has also been effectively used for prophylactic (Davidsson et al. 1989) and therapeutic benefits (Mitra et al. 1995, Sarker et al. 1998) in rotavirus diarrhoea in hospitalized children. In a recently concluded study in children with rotavirus diarrhoea in Bangladesh, we have observed a modest benefit from oral administration of immunoglobulin extracted from eggs of chicken immunized with human strains of rotavirus (Sarker et al. 2001).

Passive immunization for prevention or treatment of enteric infections generally requires relatively large amounts of antibody, particularly at the mucosal sites where antibodies are rapidly cleared. Therefore, these modalities, although proven to be effective, become expensive due to requirement of larger doses of antibodies. The other limitations of the conventional IgG antibodies include their poor stability and complex nature that limits their large-scale production. A promising solution for these problems in large-scale antibody production came, rather unexpectedly, from the nature itself- camels and llama posses an unusual type of IgG antibodies (IgG2 and IgG3) that are devoid of light chains- the "heavy chain" antibodies.

Selection of heavy chain antibody fragments In llama and camel, the "heavy chain" IgG antibodies co-exist with the "conventional" IgG (IgG1) (Hamers-Casterman et al. 1993). In contrast to conventional antibodies, the heavy chain antibodies are devoid of the light chains. Therefore, the binding domain of the heavy chain antibodies consists only of the variable domain of the heavy chain (VHH) in contrast to the binding domain of the conventional antibodies which consists of a variable domain of the heavy chain (VH) and one of the light chain (VL). The biochemical properties of llama VHH antibody fragments are superior to the Fv fragments (VH + VL) of conventional IgG antibodies. Although the VHH antibody fragments have a simple antigen binding structure with only one domain, it possesses high affinity, and is extremely thermostable (van der Linden et al., 1999). Furthermore, they are well expressed and secreted by the bakers yeast Saccharomyces cerevisiae, allowing for a large-scale cost effective production (Frenken et al., 2000). This process will make the VHH fragments an affordable ingredient for food products and will widen their availability to the general population of developing countries.

VHH as a potential food ingredient Many people in African/Arabic countries regularly consume camel milk. In 1992, it was observed that camel milk contains high titres of antibodies against rotavirus (el Agamy et al 1992).The antibody fragment in VHH batch 203027 is a fragment of those antibodies assumed to be present in camel/llama milk. Thus, the investigational product can be classified as a food ingredient As from its start in 1999, the aim of Unilever's "VHH" project was to develop an affordable food for developing countries, which "may help in reducing the risk for rotavirus infections". This type of claim fits very well into the definitions put forward by the European Union-sponsored Concerted Action on Functional Foods Science in Europe (FUFOSE) (Diplock et al 1999). The FUFOSE terminology's for 'enhanced function' (type A) and 'reduction of risk of disease' (type B) claims are now widely adapted by many national and international codes of practice, including Codex Alimentarius. It was especially developed in the 1990's to allow the delineation between functional foods from drugs. In this context, we would also like to refer to the EC Regulation No 258/97 of the European Parliament and of the Council of 27 January 1997 concerning novel foods and novel food ingredients and the EU regulation 1924/2006 on nutrition and health claims made for foods. The efficacy of VHH fragments in reducing the risk for developing rotavirus diarrhoea when supplied in a food format will be tested in an additional trial Safety of application of VHH antibody fragment Safety of oral application of VHH antibody fragment has been proven in two studies executed in the Netherlands and Bangladesh, including adult and children above the age of 6 months.

Comparison:

We will compare with the effect of VHH antibody fragment against placebo in children with proven rotavirus diarrhoea hospitalized at the ICDDR,B. This intervention will be on top of the standard treatment, including oral rehydration treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male
* Age: 6-24 months
* History of watery diarrhoea of 48 hours or less
* At least 4 liquid stools during the previous 24 hours
* No V. cholerae in a dark-field test microscopy
* Presence of rotavirus in stool as determined by ELISA
* Written informed consent for participation by respective parents/guardians

Exclusion Criteria:

* Systemic infection(s) requiring antibiotic treatment
* Severe malnutrition (W/H <-3SD)
* History of bloody diarrhoea
* Patient unwilling to comply with study protocol
* Currently participating or have participated in another clinical trial during the last 3 weeks prior to this study.

Ages: 6 Months to 24 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Diarrhoea severity (indicated by reduced stool volume) | 4-5 days
  The primary outcome measures of this study are to evaluate the efficacy of orally administered VHH batch 203027 by its ability to reduce:
  (i) diarrhoea severity (indicated by reduced stool volume) (ii) diarrhoea duration, and (iii) duration of faecal excretion of rotavirus

SECONDARY OUTCOMES:
Secondary aim: The secondary aim is to compare the influence of the passive immunisation with VHH on serum concentrations of anti-rotavirus antibody on day 4 and 21. | 4-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Shafiqul A Sarker, MD, Ph. D., Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital, Dhaka, Bangladesh

REFERENCES:
- [Derived] Sarker SA, Jakel M, Sultana S, Alam NH, Bardhan PK, Chisti MJ, Salam MA, Theis W, Hammarstrom L, Frenken LG. Anti-rotavirus protein reduces stool output in infants with diarrhea: a randomized placebo-controlled trial. Gastroenterology. 2013 Oct;145(4):740-748.e8. doi: 10.1053/j.gastro.2013.06.053. Epub 2013 Jul 2. PMID 23831050